CLINICAL TRIAL: NCT04665531
Title: Postoperative Analgesia With a Catheter Under the Erector Spinae Muscle for Videothoracoscopic Lung Surgery
Acronym: ESCAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Surgery Bitenc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120- 372/2019A
Record Dates: First submitted 2020-11-11; First posted 2020-12-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Neoplasm of Lung; Thoracic Surgery, Video-Assisted
Keywords: Anesthesia, Conduction; Regional Anesthesia; Post-operative Analgesia
MeSH Terms: conditions — Lung Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: The method of treatment is obvious and cannot be masked for care providers and investigators. Data will be non-labelled and therefore concealed before the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Erector Spinae Catheter group (Experimental): Patients in the experimental group will receive the erector spinae catheter prior the surgery and will be administered local anesthetics for 48 hours post-operatively.
  Anesthetic regimen: initial bolus of 20ml 0.5% levobupivacaine before the end of surgery. Then continually ropivacaine 0,2% 5ml/h with intermittent boluses 15ml ropivacaine 0,2% every 4h.
  Both groups will receive multimodal analgetic treatment consisting of a patient-controlled (PCA) pump with opioid analgetics and a peripherally acting analgetic metamizol on a regular basis. The PCA pump will be set to intermittent boluses of 3mg piritramide with a lock-out time 15 min and a maximal number of 6 boluses /3 hours. Patients will receive metamizol 2,5g/12hours i.v. on the day of surgery and 500-1000mg / 6 hours orally on the first and second post-operative day.
  Interventions: Procedure: Erector Spinae Catheter; Drug: Ropivacaine 0.2% Injectable Solution
- Group B - Intercostal block (Active Comparator): Patients will receive standard treatment, i.e. the multi-level intercostal block administered at the end of the surgery by the surgeon. They will receive 20ml 0,5% levobupivacaine on 6 levels of the thoracic wall according to the operative wound level.
  Both groups will receive multimodal analgetic treatment consisting of a patient-controlled (PCA) pump with opioid analgetics and a peripherally acting analgetic metamizol on a regular basis. The PCA pump will be set to intermittent boluses of 3mg piritramide with a lock-out time 15 min and a maximal number of 6 boluses /3 hours. Patients will receive metamizol 2,5g/12hours i.v. on the day of surgery and 500-1000mg / 6 hours orally on the first and second post-operative day.
  Interventions: Procedure: Intercostal block

INTERVENTIONS:
Procedure: Erector Spinae Catheter — Patients in the experimental group will receive the Erector Spinae Catheter with an initial bolus ob 20ml 0,5% levobupivacaine prior the surgery and will be administered local anesthetics for 48 hours post-operatively.
  Other Names: continuous regional analgesia
  Arms: Group A - Erector Spinae Catheter group
Procedure: Intercostal block — Patients in the comparative group will receive standard treatment, i.e. the multi-level intercostal block with 20ml 0,5% levobupivacaine administered at the end of the surgery by the surgeon.
  Other Names: Single shot regional analgesia
  Arms: Group B - Intercostal block
Drug: Ropivacaine 0.2% Injectable Solution — Patients in the experimental group will receive Ropivacaine 0,2% continous infusion of 5ml/h with boluses 15ml/4h by the Erector Spinae Catheter for 48 hours post-operatively.
  Arms: Group A - Erector Spinae Catheter group

SUMMARY:
The purpose of the research is to prove the analgesic efficacy of a novel technique in regional anaesthesia, i.e. the catheter under the erector spinae muscle (ESC). Investigators will evaluate the use of the ESC for analgesia after video-assisted thoracoscopic lung surgeries in comparison to the standard method of post-operative analgesia, which is the multiple level intercostal block given at the end of surgery by the surgeon. Investigators will compare the amount of opioid analgesics required by the patient using the patient controlled pump, the pain status in 48-hours after surgery and compare the differences between pre- and post-operative main inspiratory pressure and main expiratory pressure measurements between the two research groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* ASA (American Society of Anesthesiologists status) I-III
* Elective video-assisted thoracic surgery - lobectomy with 3 ports technique
* No contraindications for regional anesthesia

Exclusion Criteria:

* Allergy to local anesthetic
* Pregnancy, breastfeeding
* BMI>35
* Inflammation in the area of ES catheter insertion
* Inability to use the PCA pump
* Inability to execute the main inspiratory and expiratory pressure measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Demand for opioid analgetics | Continually 48 hours after surgery
  Investigators will measure the total consumption of i.v. piritramide after surgery given by the PCA (patient-controlled analgesia) pump. The PCA pump automatically marks all the drug consumption. The PCA pump will be set to a uniform protocol: piritramide 1mg/ml; flow 0ml/h, bolus 3ml, lockout time 15 min, max 4 boluses / hour.
Difference in pre- and post-operative respiratory muscle fitness | First postoperative day
  Investigators will compare the change between pre- and post-operative main inspiratory pressure and main expiratory pressure measurements between the two research groups.
Difference in pre- and post-operative respiratory muscle fitness | Second postoperative day
  Investigators will compare the change between pre- and post-operative main inspiratory pressure and main expiratory pressure measurements between the two research groups.

SECONDARY OUTCOMES:
Subjective pain score | Every hour in the 48 hours post surgery.
  Investigators will measure subjective perception of pain with the nubmering rating score (NRS) scoring system at resting and coughing. The NRS scoring system is a numerical scale from 0-10, with 0 being no pain and 10 the strongest pain imaginable. Patients will assess their pain with the help of analogue scale with colours and faces by each number representing different NRS pain levels.

OTHER OUTCOMES:
Number of patients with late post-operative complications | 2 months
  Investigators will follow up the patients in 4 and 12 weeks after surgery for possible complications. The complications will be read from the follow up documentation in observed patient files. Investigators will search for complications such as arrhythmias, lung or wound infections, lethalities or other unexpected complications.

CONTACTS AND LOCATIONS:
Overall Officials: Polona Gams, Principal Investigator — Surgery Bitenc
Locations (1):
- Surgery Bitenc, Golnik, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Beverly A, Kaye AD, Ljungqvist O, Urman RD. Essential Elements of Multimodal Analgesia in Enhanced Recovery After Surgery (ERAS) Guidelines. Anesthesiol Clin. 2017 Jun;35(2):e115-e143. doi: 10.1016/j.anclin.2017.01.018. PMID 28526156
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Bialka S, Copik M, Daszkiewicz A, Rivas E, Ruetzler K, Szarpak L, Misiolek H. Comparison of different methods of postoperative analgesia after thoracotomy-a randomized controlled trial. J Thorac Dis. 2018 Aug;10(8):4874-4882. doi: 10.21037/jtd.2018.07.88. PMID 30233861
- [Background] Ahmed Z, Samad K, Ullah H. Role of intercostal nerve block in reducing postoperative pain following video-assisted thoracoscopy: A randomized controlled trial. Saudi J Anaesth. 2017 Jan-Mar;11(1):54-57. doi: 10.4103/1658-354X.197342. PMID 28217054
- [Background] D'Ercole F, Arora H, Kumar PA. Paravertebral Block for Thoracic Surgery. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):915-927. doi: 10.1053/j.jvca.2017.10.003. Epub 2017 Oct 4. PMID 29169795
- [Background] Ilfeld BM, Gabriel RA. Basal infusion versus intermittent boluses for perineural catheters: should we take the 'continuous' out of 'continuous peripheral nerve blocks'? Reg Anesth Pain Med. 2019 Mar;44(3):285-286. doi: 10.1136/rapm-2018-100262. Epub 2019 Jan 13. No abstract available. PMID 30636717
- [Background] Kamiyoshihara M, Nagashima T, Ibe T, Atsumi J, Shimizu K, Takeyoshi I. Is epidural analgesia necessary after video-assisted thoracoscopic lobectomy? Asian Cardiovasc Thorac Ann. 2010 Oct;18(5):464-8. doi: 10.1177/0218492310381817. PMID 20947601
- [Background] Krebs ED, Mehaffey JH, Sarosiek BM, Blank RS, Lau CL, Martin LW. Is less really more? Reexamining video-assisted thoracoscopic versus open lobectomy in the setting of an enhanced recovery protocol. J Thorac Cardiovasc Surg. 2020 Jan;159(1):284-294.e1. doi: 10.1016/j.jtcvs.2019.08.036. Epub 2019 Sep 13. PMID 31610965
- [Background] Adhikary SD, Pruett A, Forero M, Thiruvenkatarajan V. Erector spinae plane block as an alternative to epidural analgesia for post-operative analgesia following video-assisted thoracoscopic surgery: A case study and a literature review on the spread of local anaesthetic in the erector spinae plane. Indian J Anaesth. 2018 Jan;62(1):75-78. doi: 10.4103/ija.IJA_693_17. PMID 29416155
- [Background] Hong B, Bang S, Chung W, Yoo S, Chung J, Kim S. Multimodal analgesia with multiple intermittent doses of erector spinae plane block through a catheter after total mastectomy: a retrospective observational study. Korean J Pain. 2019 Jul 1;32(3):206-214. doi: 10.3344/kjp.2019.32.3.206. PMID 31257829